CLINICAL TRIAL: NCT04924348
Title: WALANT (Wide Awake Local Anaesthesia With No Tourniquet) Procedure in Carpal Tunnel Release: a Prospective Randomized Study
Brief Title: WALANT Procedure in Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WALANT; 2020-A00446-33 (Other: ANSM)
Record Dates: First submitted 2021-05-24; First posted 2021-06-14 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Carpal Tunnel; Median Nerve Neuralgia; Anesthesia, Local
MeSH Terms: conditions — Median Neuropathy

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, therapeutic, comparative, randomized controlled open-label, non-inferiority, single-center, national study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WALANT procedure (Experimental): Local anesthesia of the WALANT type
  Interventions: Procedure: Experimental: WALANT procedure
- Axial ALR (Active Comparator): Axillary loco-regional anesthesia
  Interventions: Procedure: Active Comparator: Axial ALR
- Truncal ALR (Active Comparator): Truncal loco-regional anesthesia
  Interventions: Procedure: Active Comparator: Truncal ALR

INTERVENTIONS:
Procedure: Experimental: WALANT procedure — The WALANT technique, performed under ultrasound, includes two punctures.
  * The first is a puncture through a medial approach above the wrist and includes two injections. A first subcutaneous injection reproducing a bar above the wrist flexion line, and a second injection above the median nerve. The volumes injected vary from 8 to 10 milliliters (ml).
  * The second puncture is performed at the base of the palmar surface of the hand and consists of a 10 ml subcutaneous injection of the local anesthetic in order to take advantage of the vasoconstrictive effects of adrenaline, thus allowing the surgical procedure to be performed without a pneumatic tourniquet.
  Arms: WALANT procedure
Procedure: Active Comparator: Axial ALR — The anesthetic protocol in the axillary block consists of performing a puncture, using a needle (50 mm 22G with a short bevel), under the armpit at the level of the axillary hollow after skin disinfection. This puncture, performed under ultrasound, allows the injection of the local anesthetic around the median, radial, ulnar and musculocutaneous nerves. The volume injected per nerve can vary from 5 to 8 ml depending on the visual appreciation during the injection.
  Arms: Axial ALR
Procedure: Active Comparator: Truncal ALR — The anesthetic protocol in truncal block consists in injecting the local anesthetic around the median and ulnar nerves by a puncture performed at the elbow or forearm (depending on the practitioner's experience). The volumes injected remain the same and the puncture is also performed under ultrasound guidance. Additional local anesthesia is administered by injecting an additional 5 ml above the wrist flexion line to block the sensory territory of the musculocutaneous nerve.
  Arms: Truncal ALR

SUMMARY:
The possible benefits expected from the use of the WALANT procedure are a decrease in intraoperative pain at the surgical site, a decrease in hospitalization time, and a decrease in the time required to lift the anesthesia postoperatively.

The risks identified are those inherent to each type of anesthesia (WALANT or traditional ALR), as encountered in current practice, and are therefore not specific to the study: risks related to the local anesthetic agent or risks related to the puncture procedure.

The main objective is to determine whether the patient's intraoperative pain at the surgical site is less after a WALANT procedure compared to a traditional ALR procedure (axillary or trunk).

DETAILED DESCRIPTION:
Median nerve neurolysis at the carpal tunnel is one of the most performed procedures in the world. The use of loco-regional anesthesia (LRA) is common practice for this surgery, especially since the use of ultrasound guidance, which allows visualization of the nerves and control of the injection of anesthetic products, makes it a safe technique. The nerve blocks most commonly used in hand surgery are axillary blocks and truncal blocks. The choice between these two techniques, which are equivalent in terms of effectiveness and duration of anesthesia, depends in practice on the habits of each practitioner. As the use of a pneumatic tourniquet during the operation is systematic, the axillary block, by anaesthetizing the whole arm, avoids the discomfort described by some patients when using a tourniquet. For others, the discomfort is related to the sensation of a "dead arm" with a duration of anesthesia of several hours, which the truncular block makes it possible to avoid.

Recently, an alternative to traditional LRA by local anesthesia without tourniquet and without sedation (WALANT procedure: Wide Awake Local Anesthesia with No Tourniquet) has been described. Several studies show the efficacy and safety of this procedure, which is already used in current practice.

However, to date, there is no comparative study evaluating the effectiveness of the WALANT procedure compared to traditional hand surgery techniques for carpal tunnel, neither published nor in progress. This is the purpose of this study.

The WALANT technique, performed under ultrasound, includes two punctures.

* The first is a puncture through a medial approach above the wrist and includes two injections. A first subcutaneous injection reproducing a bar above the wrist flexion line, and a second injection above the median nerve. The volumes injected vary from 8 to 10 milliliters (ml).
* The second puncture is performed at the base of the palmar surface of the hand and consists of a 10 ml subcutaneous injection of the local anesthetic in order to take advantage of the vasoconstrictive effects of adrenaline, thus allowing the surgical procedure to be performed without a pneumatic tourniquet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient over 18 years of age
* Membership in a mandatory health insurance plan
* Patient treated for a first median nerve liberation surgery at the carpal tunnel
* Patient having been informed of the study and having given informed consent
* French-speaking patient

Exclusion Criteria:

* Surgical revision
* Contraindication(s) to loco-regional anesthesia :

  1. Coagulation disorder or ongoing anticoagulant therapy
  2. Existing peripheral neuropathy
  3. Amide-type AL allergy
* Pregnant or breastfeeding women
* Inability to undergo the medical follow-up of the study for geographical, social or psychological reasons
* Patients under legal protection
* Patients under the influence of drugs that may interfere with the anesthetic techniques under study (cocaine, cannabis, etc. as judged by the investigator)
* Inclusion of the subject in another research protocol during this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of the patient's pain intraoperatively at the surgical site. | Within 24 hours after intervention
  Evaluation of the patient's pain, at the level of the operative site by a visual analog scale from 0 to 10 where 0 equals to "No Pain" and 10 equals to "Extremely severe pain".

SECONDARY OUTCOMES:
Visual Analog Scale for intraoperative pain at the surgical site | intraoperative
  The assessment of pain at the surgical site will be evaluated using a 10-point visual analog scale score from 0 to 10 where 0 equals to "No Pain" and 10 equals to "Extremely severe pain"
Satisfaction scores | Within 24 hours after intervention
  Satisfaction scores according to the forms provided in the appendices of the anaesthetist and the surgeon
Satisfaction scores | One day after intervention
  Satisfaction scores according to the forms provided in the appendices of the patient
Assessment of the patient's overall pain after surgery | One day after intervention
  Assessment of the patient's overall pain after surgery using a numerical scale (EN) from 0 to 10 where 0 equals to "No Pain" and 10 equals to "Extremely severe pain"
Assessment of the patient's overall pain after surgery | One month after intervention
  Assessment of the patient's overall pain after surgery using a numerical scale (EN) from 0 to 10 where 0 equals to "No Pain" and 10 equals to "Extremely severe pain"
Assessment of the patient's overall pain after surgery | Three months after intervention
  Assessment of the patient's overall pain after surgery using a numerical scale (EN) from 0 to 10 where 0 equals to "No Pain" and 10 equals to "Extremely severe pain"
Assessment of the patient's overall pain after surgery | Six months after intervention
  Assessment of the patient's overall pain after surgery using a numerical scale (EN) from 0 to 10 where 0 equals to "No Pain" and 10 equals to "Extremely severe pain"
Evaluation of the return to work after surgery | Within 24 hours after intervention
  Evaluation thanks to the Quick-DASH Questionnaire from 0 to 100 where 0 equals to "No disability" and 100 equals to "Most severe disability and reduced function"
Evaluation of the return to work after surgery | One month after intervention
  Evaluation thanks to the Quick-DASH Questionnaire from 0 to 100 where 0 equals to "No disability" and 100 equals to "Most severe disability and reduced function"
Evaluation of the return to work after surgery | Three months after intervention
  Evaluation thanks to the Quick-DASH Questionnaire from 0 to 100 where 0 equals to "No disability" and 100 equals to "Most severe disability and reduced function"
Evaluation of the return to work after surgery | Six months after intervention
  Evaluation thanks to the Quick-DASH Questionnaire from 0 to 100 where 0 equals to "No disability" and 100 equals to "Most severe disability and reduced function"
Evaluation of the quality of life | Baseline (Before the anesthesia)
  Evaluation thanks to the SF-36 from 0 to 100 where 0 equals to "Poor Health" and 100 equals to "Good Health"
Evaluation of the quality of life | One month after intervention
  Evaluation thanks to the SF-36 from 0 to 100 where 0 equals to "Poor Health" and 100 equals to "Good Health"
Evaluation of the quality of life | Three months after intervention
  Evaluation thanks to the SF-36 from 0 to 100 where 0 equals to "Poor Health" and 100 equals to "Good Health"
Evaluation of the quality of life | Six months after intervention
  Evaluation thanks to the SF-36 from 0 to 100 where 0 equals to "Poor Health" and 100 equals to "Good Health"
Evaluation of the use of analgesics in the postoperative situation | One day after intervention
  The use of analgesics will be collected until D+1 by defining the following levels of analgesic intake:
  * Level I: use of a paracetamol-type analgesic, up to 4 g/day
  * Level II: use of another type of analgesic (Tramadol or Lamaline®)
Evaluation of the failure rates of different anesthesia procedures. | Within 24 hours after intervention
  The following were considered procedural failures: need for intravenous sedation for all 3 groups, need to inflate the tourniquet (applied as a preventive measure) for the WALANT group only.
Evaluation of the operative time. | During surgery
  Operating time defined as the time from skin incision to skin closure (in minutes)
Evaluation of the hospitalization length. | Within 24 hours after intervention
  Hospitalization length defined as the time from the patient's admission to the end of the hospitalization (in hours)
Evaluation of the time to release of anesthesia. | Within 24 hours after intervention
  Time to release of anesthesia defined as the time from the placement of anesthesia to the release of motor (ability to clench/unclench the hand) and sensory (disappearance of tingling) anesthesia
Evaluation of the safety of different types of anesthesia. | One month after intervention
  Collection of postoperative adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Flore-Anne LECOQ, MD, Principal Investigator — Institut de la Main Nantes Atlantique
Locations (1):
- Institut de la main Nantes Atlantique, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lalonde DH. Conceptual origins, current practice, and views of wide awake hand surgery. J Hand Surg Eur Vol. 2017 Nov;42(9):886-895. doi: 10.1177/1753193417728427. Epub 2017 Sep 8. PMID 28886668
- [Background] Tulipan JE, Kim N, Abboudi J, Jones C, Liss F, Kirkpatrick W, Rivlin M, Wang ML, Matzon J, Ilyas AM. Open Carpal Tunnel Release Outcomes: Performed Wide Awake versus with Sedation. J Hand Microsurg. 2017 Aug;9(2):74-79. doi: 10.1055/s-0037-1603200. Epub 2017 May 22. PMID 28867906
- [Background] Lalonde D, Martin A. Tumescent local anesthesia for hand surgery: improved results, cost effectiveness, and wide-awake patient satisfaction. Arch Plast Surg. 2014 Jul;41(4):312-6. doi: 10.5999/aps.2014.41.4.312. Epub 2014 Jul 15. PMID 25075350
- [Background] Steiner MM, Calandruccio JH. Use of Wide-awake Local Anesthesia No Tourniquet in Hand and Wrist Surgery. Orthop Clin North Am. 2018 Jan;49(1):63-68. doi: 10.1016/j.ocl.2017.08.008. PMID 29145985
- [Background] Wright J, MacNeill AL, Mayich DJ. A prospective comparison of wide-awake local anesthesia and general anesthesia for forefoot surgery. Foot Ankle Surg. 2019 Apr;25(2):211-214. doi: 10.1016/j.fas.2017.10.015. Epub 2017 Nov 6. PMID 29409279
- [Background] Fayad F, Lefevre-Colau MM, Gautheron V, Mace Y, Fermanian J, Mayoux-Benhamou A, Roren A, Rannou F, Roby-Brami A, Revel M, Poiraudeau S. Reliability, validity and responsiveness of the French version of the questionnaire Quick Disability of the Arm, Shoulder and Hand in shoulder disorders. Man Ther. 2009 Apr;14(2):206-12. doi: 10.1016/j.math.2008.01.013. Epub 2008 Apr 23. PMID 18436467
- [Background] Estebe JP, Gentili ME, Langlois G, Mouilleron P, Bernard F, Ecoffey C. Lidocaine priming reduces tourniquet pain during intravenous regional anesthesia: A preliminary study. Reg Anesth Pain Med. 2003 Mar-Apr;28(2):120-3. doi: 10.1053/rapm.2003.50123. PMID 12677622
- See also: Points to consider on multiplicity issues in clinical trials, EMEA, 2002 — https://www.ema.europa.eu/en/documents/scientific-guideline/points-consider-multiplicity-issues-clinical-trials_en.pdf